# Massachusetts-wide study of the incidence of ATrial fibRIllation and stroke occurring after discharge from Cardiac Surgery (MATRICeS)

Principal Investigator:

Simon C. Body, MBChB, MPH, FAHA <a href="mailto:sbody@bwh.harvard.edu">sbody@bwh.harvard.edu</a>

Co-Investigators:

J. Daniel Muehlschlegel, MD, MMSc, FAHA <u>imuehlschlegel@bwh.harvard.edu</u>

Bala Subrama@bidmc.harvard.edu bsubrama@bidmc.harvard.edu

Xinling (Claire) Xu, PhD <a href="mailto:xxu20@bwh.harvard.edu">xxu20@bwh.harvard.edu</a>

Abdallah Alameddine, M.D. <u>akalameddine@gmail.com</u>

Vladimir Birjiniuk, M.D. <u>vbirjini@mah.harvard.edu</u>

Frederick Y. Chen, M.D. fchen1@tuftsmedicalcenter.org

Iraklis Gerogiannis, M.D. <a href="mailto:gerogiannisi@southcoast.org">gerogiannisi@southcoast.org</a>

Tsuyoshi Kaneko, M.D. <u>tkaneko2@bwh.harvard.edu</u>

Kamal Khabbaz@bidmc.harvard.edu kkhabbaz@bidmc.harvard.edu

Paul Pirundini, M.D. <a href="mailto:ppirundini@capecodhealth.org">ppirundini@capecodhealth.org</a>

Thoralf M. Sundt, M.D. <u>tsundt@mgh.harvard.edu</u>

Jennifer Walker, M.D. jennifer.walker@umassmemorial.org

IRB Number: 2017P002261 Partners HealthCare IRB.

**Authors of the Statistical Analysis Plan:** 

Simon C. Body, MBChB, MPH, FAHA

Xinling (Claire) Xu, PhD

Initial version date: 2/15/2018

| Amendment 1: |
|-----------------------|
| Amended version date: |
| Changes in Amendment: |
| Amendment 2: |
| Amended version date: |
| Changes in Amendment: |
| Amendment 3: |
| Amended version date: |
| Changes in Amendment: |
| Amendment 4: |
| Amended version date: |
| Changes in Amendment: |
| Amendment 5: |
| Amended version date: |
| Changes in Amendment: |

# **Table of Contents**

| <u>1</u> | INTRODUCTION | <u>5</u> |
|---|---|---|
| 1.1 | Study Introduction | 5 |
| 1.2 | | |
| 2 | STUDY SUMMARY AND AIMS | 6 |
| <u> </u> | 51001 30MMART AND AIMS | <u></u> |
| | Course Province | , |
| 2.1 | | |
| <ul><li>2.2</li><li>2.3</li></ul> | | |
| 2.3<br>2.4 | | |
| 2.4 | SECONDARY AIMS | / |
| <u>3</u> | STUDY ENDPOINTS AND COVARIATES | <u>7</u> |
| 3.1 | DEFINITIONS OF STUDY ENDPOINTS | |
| 3.2 | DEFINITIONS OF COVARIATES | |
| 3.3 | MODIFICATIONS OR DERIVATIONS OF STANDARD VARIABLES | |
| 3.4 | UNRELATED OUTCOMES | 8 |
| <u>4</u> | ESTIMATION OF ACCESSIBLE EFFECT SIZE | <u>8</u> |
| 5 | DATA SOURCES | 8 |
| _ | | |
| 6 | STUDY POPULATIONS | Я |
| <u> </u> | 510D11 OF CEATIONS | ······ |
| 6.1 | Inclusion Criteria | 0 |
| 6.1 | EXCLUSION CRITERIA | |
| 6.2<br>6.3 | SUBGROUPS | |
| 6.4 | DESCRIPTION OF PARTICIPANTS | |
| <b>0.</b> 4 | DESCRIPTION OF PARTICIPANTS | |
| _ | CTATICTICAL ANALYCEC | _ |
| <u>/</u> | STATISTICAL ANALYSES | <u></u> 9 |
| 7.1 | | |
| 7.1. | | |
| 7.1. | | |
| | POOLING OF SITES | |
| 7.3 | | |
| 7.4 | | |
| 7.4.<br>7.4 | 1 ADJUSTMENTS FOR COVARIATES | |
| 7.4. | Z IVIULTIPLE CUMPARISONS | 11 |

| 7.4.3 | B Examination of Subgroups | 11 |
|---|---|---|
| 7.4.4 | CORRELATED DATA, BIAS, CONFOUNDING AND INTERACTIONS | 11 |
| 7.4.5 | SUBGROUP ANALYSES | 11 |
| 7.5 | POST-HOC (DATA DRIVEN) ANALYSES: | 11 |
| 7.6 | SENSITIVITY ANALYSES | 12 |
| <u>8</u> <u>A</u> | APPENDIX: STUDY ADMINISTRATION | 13 |
| 8.1 | CONFIDENTIALITY | 13 |
| 8.2 | RECORDS RETENTION | 13 |
| 8.3 | INFORMED CONSENT/ASSENT AND HIPAA AUTHORIZATION | 13 |
| 9 <u>A</u> | APPENDIX: DATA TO BE OBTAINED FROM MASSACHUSETTS CARDIAC SURGICAL PROGRAMS | 14 |
| <u>10</u> | APPENDIX: CHIA-SOURCED VARIABLE DEFINITIONS AND ABSTRACTION | 22 |
| <u>11</u> | APPENDIX: PROPOSED TIMELINE | 23 |
| <u>12</u> | APPENDIX: SHELL TABLES AND FIGURES | 24 |
| 12.1 | Tables | 24 |
| 12.2 | FIGURES | 24 |
| <u>13</u> | APPENDIX: STROBE CRITERIA | 33 |
| 14 | APPENDIX: REFERENCES | 35 |

#### 1 INTRODUCTION

This Statistical Analysis Plan codifies the analysis of a retrospective research study that has been previously reviewed and approved (2017P002261) by the Partners HealthCare Institutional Review Board (IRB) and will be conducted in accordance with all applicable human subjects' research requirements and applicable federal regulations.

#### 1.1 Study Introduction

Briefly, this study examines the occurrence and neurological consequences of atrial fibrillation, occurring after discharge to home or rehab after cardiac surgery. The study examines patients who underwent cardiac surgery at Cardiac Surgical Programs in Massachusetts between 1/1/2012 and 12/31/2016, with a follow-up period that extends to 12/31/2017.

Detailed data will be obtained from individual Programs that encompasses preoperative medical history, the operative period including details about the operation and also the post-operative period until discharge from hospital. Information about the post-hospital discharge course for individual patients will be obtained from the Massachusetts Center for Health Information and Analysis (CHIA) (<a href="https://www.mass.gov/orgs/center-for-health-information-and-analysis">https://www.mass.gov/orgs/center-for-health-information-and-analysis</a>). CHIA collects detailed financial and patient-level data from Massachusetts payers and providers, and makes it available to researchers.

#### 1.2 Background Literature

Atrial fibrillation (AF) is the most common cardiac arrhythmia and frequently presents in association with mitral, other valvular and coronary artery disease, notably in the presence of poorer left ventricular function (1,2). Preoperative AF is reported commonly in patients undergoing cardiac surgery, with an incidence of 10-20% (2-8). Even if treated, preoperative AF is associated with a higher incidence of inhospital postoperative AF, stroke, other cardiac morbidity and mortality (2,6,9-11).

Conventional management of postoperative AF assumes that it results from self-limited causes, such as postoperative pericarditis, surgical stress, and sympathetic stimulation in patients underlying heart disease that can be treated with short-term antiarrhythmics, heart rate reduction, anti-coagulants and anti-platelet agents. However, it is well-known that AF in the immediate postoperative period is associated with increased risk of post-discharge AF and stroke. Observed incidences range widely (3-25%) depending principally on the duration of follow-up and the mode of monitoring (12-14). These studies did not use continuous ECG monitoring to detect AF recurrence, and therefore may have underestimated the incidence of AF by missing asymptomatic AF. Using continuous ECG monitoring the incidence of at least one electrocardiographic episode of AF lasting longer than six minutes is much higher; 60% over the entire follow-up period and 39% occurring more than 3-months after surgery (15).

Thromboembolic stroke is a major preventable cause of morbidity and mortality in patients with post-operative AF (16-18). Studies have demonstrated a risk-unadjusted two to ten-fold increase in embolic events and a threefold increased risk of cardiac death in patients with postoperative AF (12,19,20).

The efficacy of concomitant AF ablation in patients undergoing cardiac surgery, measured as freedom from AF and quality of life, and safety measured as freedom from morbidity and mortality, has been well demonstrated (21-29), especially after mitral valve surgery. Observational studies with large sample sizes and longer follow-up have demonstrated improved survival after surgical ablation in normal sinus rhythm (30-33). Yet the implementation of AF ablation and stroke reduction procedures, while increasing (34,35), remains relatively low in the US (33). This is despite guidelines from National and International Societies (36-39) that support use of these procedures. Concerns voiced about concomitant AF ablation or stroke reduction surgery include increased operative time and complexity, perceived operative risk of the procedures (40), and increased risk of atrio-ventricular block requiring pacemaker insertion (21,34,35,41,42).

#### 2 STUDY SUMMARY AND AIMS

The purpose of this study is to determine the incidence, risk factors and adverse events consequent upon atrial fibrillation after cardiac surgery, as well as the association between prior atrial fibrillation and postoperative atrial fibrillation. The study uses information from local Cardiac Surgical Programs to describe the preoperative medical state and immediate post-operative state. Additionally, information from the post-discharge period will be provided by CHIA, by matching the two sources of information using HIPAA-waived data such as medical record number, date of birth, gender and last name. Once matched, the data are stripped of identifiers.

#### 2.1 Study Design:

We will employ a retrospective cohort design, examining patients who underwent cardiac surgery at Cardiac Surgical Programs in Massachusetts between 1/1/2012 and 12/31/2016, with a follow-up period that extends to 12/31/2017. The study examines the risk factors and incidence of post-operative atrial fibrillation, stroke and other focal neurological events after discharge from hospital.

#### 2.2 Study Population and Sites

The study will examine the medical records of patients who underwent cardiac surgery in Massachusetts between 1/1/2012 to 12/31/2016. It is estimated that ~50,000 patients are eligible for inclusion in this study. The evaluable sample size is derived from a sample of convenience from the following Institutions.

Baystate Medical Center, Springfield, MA
Beth Israel Deaconess Medical Center, Boston, MA
Brigham and Women's Hospital, Boston, MA
Cape Cod Hospital, Hyannis, MA
SouthCoast Health, Fall River, MA
Massachusetts General Hospital, Boston, MA
Mount Auburn Hospital, Cambridge, MA
UMass Memorial Medical Center-University, Worcester, MA

Tufts Medical Center, Boston, MA

#### 2.3 Primary Aims

The Primary Aims of this study are to determine:

- The risk factors, which includes the main risk factor preoperative atrial fibrillation, for postoperative atrial fibrillation occurring after discharge from hospital in patients who underwent cardiac surgery during admission.
- 2. The risk factors, which includes the main risk factor preoperative atrial fibrillation, for stroke or other focal neurologic event occurring after discharge from hospital in patients who underwent cardiac surgery during admission.

#### 2.4 Secondary Aims

The Secondary Aims of this study are to determine:

- 1. The frequency of, and treatments for, atrial fibrillation occurring after discharge from hospital in patients who underwent cardiac surgery during admission.
- 2. The frequency of stroke or other focal neurologic event occurring after discharge from hospital in patients who underwent cardiac surgery during admission
- 3. The incidence of all-cause and stroke-related mortality after cardiac surgery.

#### 3 STUDY ENDPOINTS AND COVARIATES

#### 3.1 Definitions of Study Endpoints

- 1. Postoperative atrial fibrillation occurring after discharge from hospital
- 2. Stroke or other focal neurologic event occurring after discharge from hospital
- 3. All-cause mortality
- 4. Stroke-related mortality

#### 3.2 Definitions of Covariates

Data derived from individual sites will use definitions from the Society of Thoracic Surgeons Adult Cardiac Surgery Database versions 2.7.3 and 2.8.2 (43,44).

#### 3.3 Modifications or derivations of standard variables

Hospital admissions will be defined using continuous in-patient stays (CIS) which combine data from each event within hospital, which includes within hospital transfers. Diagnostic subgroups will be defined using the code recorded for the main diagnosis for the first event within a CIS. The ninth

International Classification of Disease codes (ICD-9) codes will be used to define the specific conditions of interest.

#### 3.4 Unrelated outcomes

Un-related events such as upper or lower limb fracture and xxx will be used as negative controls.

Unrelated adverse events (such as upper or lower limb fracture), which are known not to be caused by prior AF will be used as the composite negative control outcome to examine whether there is unmeasured confounders of the prior AF-postoperative AF association. An observed association between prior-AF and the negative control outcome will reflect the existence of unmeasured confounders. In such cases, these unmeasured confounders will also affect the true prior AF-postoperative AF association (45). When such unmeasured confounding effect is detected, we will provide an adjusted estimate for the hazard ratio of first postoperative AF using an indirect approach (46)

#### 4 ESTIMATION OF ACCESSIBLE EFFECT SIZE

This will be a retrospective cohort study. Patients will be included in the study based on the inclusion and exclusion criteria. All statistical tests will be two-sided and the statistical significance level will be set at 0.05 unless otherwise stated. Assuming 50,000 patients will be included in the analysis, among which 4000 (8%) have prior AF, we will have 80% power to detect a Cohen's effect size of 0.046 at the 0.05 significance level. If 25% of the patients who do not have prior AF have postoperative AF, a Cohen's effect size of 0.046 is corresponding to a 2% difference in the incidence of postoperative AF.

#### 5 DATA SOURCES

#### 6 STUDY POPULATIONS

#### **6.1** Inclusion Criteria

Inclusion criteria for this study are patients who undergo surgical procedures that include coronary artery bypass graft surgery, aortic valve surgery or mitral valve surgery and other valvular surgical procedures.

#### 6.2 Exclusion Criteria

Exclusion criteria for this study are:

Preoperative status

Prior AF ablation or pulmonary vein isolation procedure of any type Prior LA occlusion or ablation procedure of any type

Surgical procedure

MAZE or other procedure for the treatment or prevention of AF

Ventricular assist device
Heart transplantation
Bacterial endocarditis
Cardiac trauma
Cardiac tumor
Ventricular septal defect repair
Left ventricular aneurysm repair
Pulmonary thromboendarterectomy
Surgical ventricular restoration

#### 6.3 Subgroups

Subgroups may be used in secondary analyses.

#### 6.4 Description of participants

The study participants will be presented as per the CONSORT recommendations (Figure 1). The baseline characteristics will be presented (Table 1). Including:

Demographic characteristics (e.g., age, sex, socioeconomic status)

Baseline exposure characteristics (e.g., smoke exposure)

Baseline disease characteristics

Table 2 (Appendix) will describe the baseline characteristics of the study group comparing patients with post-discharge AF, compared to those without.

Baseline values of primary and/or secondary outcome variables

#### 7 STATISTICAL ANALYSES

#### 7.1 General

Baseline and demographic characteristics will be summarized using descriptive statistics (means, standard deviations or median, interquartile ranges for continuous variables such as age and percentages for categorical variables such as race and ethnicity. When deemed appropriate, they will be compared using Chi-square test, Fisher's exact test, two-sample t test, and Wilcoxon rank-sum test between groups. For each binary outcome we will report odds ratios with 95% confidence intervals and give a two-sided p-value for statistical significance. For analysis of the pre-specified subgroups (primary outcome only) we will report relative risks with 99% confidence intervals with two-sided p-value.

#### 7.1.1 Primary Aims

The standard Cox proportional hazards model will be used to model time to first atrial fibrillation occurrence and time to first stroke or other focal neurologic event, after discharge from hospital,

respectively. The potential risk factors included will be selected based on their univariate association with first event status, as well as clinical significance. Hazard ratios with 95% confidence intervals will be reported with a two-sided p-value for statistical significance. The proportional hazard assumption will be evaluated using graphical tool, and by including time dependent covariate terms.

Since there might be repeated occurrences of atrial fibrillation and stroke or other focal neurologic event for each patient, we will use the Andersen-Gill (AG) model and the Prentice, Williams and Peterson (PWP) models to analyze recurrent events data. The AG model is suitable when the interest is in the overall effect on the intensity of the occurrence of a recurrent event. The PWP models allow us to evaluate the effects of risk factors for the kth event after discharge from hospital, as well as the effects of risk factors for the kth event since the time from the previous event (47). Hazard ratios with 95% confidence intervals will be reported with a two-sided p-value for statistical significance. For time-to-event data analyses, death will be considered a censoring event.

#### 7.1.2 Secondary Aims

Means and standard deviations will be estimated for count outcomes. We will report the two-sided p-value for statistical significance of the difference in means of count outcomes.

The frequencies of atrial fibrillation and stroke or other focal neurologic event will be modeled with Poisson regression with the length of follow-up time as the offset. Potential risk factors included in this model will be selected based on univariate test results, as well as clinical significance. Logistic regression will be used to model the incidence of all-cause and stroke-related mortality after cardiac surgery, respectively.

#### 7.2 Pooling of Sites

The data will be pooled across all participating sites. In logistic and Cox proportional hazards models, site will be treated as a random effect.

#### 7.3 Methods for Handling Missing Data

The frequency and percentage of missing values for each variable will be collected, analyzed and reported. If there are missing values for the outcome variable(s), individual patients will be excluded. Highly incomplete covariates (>33% of observations missing) will be excluded from analyses. If missing values are Missing Completely At Random (MCAR), exclusion of patients with missing observations will be considered. If missing values are Missing At Random (MAR) or not at random (MNAR), multiple imputation will be performed. Missing values, selection or exclusion of observations and variables and handling of missing values in the statistical analysis will be describes carefully and sensitivity analysis will be provided (48-51)

#### 7.4 Statistical Analytical Issues

#### 7.4.1 Adjustments for covariates

There will be covariate adjustment in the primary analysis.

#### 7.4.2 Multiple Comparisons

There will be no adjustment for multiple comparisons. We will report 99% confidence intervals for subgroup analyses of the primary outcome.

#### 7.4.3 Examination of Subgroups

To determine if all subgroups experience similar treatment effects or if there are subgroups that behaved differently. We will report odds ratios with 99% confidence intervals for the primary outcome by the following subgroups, with/without prior atrial fibrillation before surgery, and with/without atrial fibrillation when discharged. We will conduct a test of homogeneity of effects across the subgroups and report a P value. Unless there is strong evidence against the null hypothesis of homogeneity of effects (i.e. p<0.001) the overall odds ratios will be considered as the most reliable guide to the approximate relative risks in all subgroups.

#### 7.4.4 Correlated data, bias, confounding and interactions.

Collinearity between risk factors will be evaluated with Variance Inflation Factors (VIF) or generalized VIF. Risk factors with high VIF (>2.5) will be excluded in the models.

#### 7.4.5 Subgroup analyses

Subgroup analyses will be performed as post-hoc analyses to determine if all subgroups experience similar treatment effects or if there are subgroups that behaved differently. The methods will be determined based on:

- Pre-specify subgroups that will be analyzed. Consider subgroups defined by:
  - Baseline values of outcome variables
  - Different types of baseline disease status (e.g., prior atrial fibrillation history)
  - Different levels of key prior exposures (e.g., smoking status/exposure, atrial fibrillation status at discharge)
- Pre-specify how the results will be interpreted:
  - We expect to see that the effects of risk factors will be in the same direction with different intensities. If we are able to identify certain subgroups that are significantly different from others, we will report the results with suggestions for future studies.

#### 7.5 Post-hoc (data driven) analyses:

Post-hoc data driven analyses are allowed after the following are undertaken.

- (a) Document which analyses were conducted after the results for the Primary and Secondary Aims are analyzed.
- (b) Document the rationale for these analyses.
- (c) Pre-specify their interpretation in the context of the primary and secondary results and their impact on the overall trial conclusions.

#### 7.6 Sensitivity Analyses

The negative control outcome analysis mentioned in section 3.4 will be part of the sensitivity analyses, which evaluates whether there is unmeasured confounding effect in the prior AF-postoperative AF association. A similar analysis will be performed for stroke, and all-cause mortality. Additionally, we will report E-values for the associations from these models. The E-value is defined as the minimum strength of association, that an unmeasured confounder would need to have with both the exposure and the outcome to fully explain away a specific exposure-outcome association, conditional on the measured covariates

When patient characteristics are significantly different between the prior AF group and non-prior AF group, stratified proportional hazard models with two sets of coefficients will be fitted, and the effects of risk factors will be evaluated. Consistency of the two sets of coefficients would reflect the imbalance of baseline variables is negligible, and one final model will be reported. For the analysis of recurrent data, consistency of the results from AG and PWP models will be monitored.

#### 8 APPENDIX: STUDY ADMINISTRATION

#### 8.1 Confidentiality

Data will be stored on encrypted hard drives and backed up to secure Partners-maintained storage within the Partners firewall. Secure transfer methods will be used. Final results will be reported in aggregate with no individually identifying data.

Linkage is done on a stand-alone PC which is not used by the analysts. The linkage process uses only temporary data sets that are immediately removed once the program has completed. The final analytic data set does not contain any patient names, addresses, or social security numbers. It also does not contain any CHIA case mix data fields.

#### 8.2 Records Retention

We anticipate follow-on studies in the field that can be performed with this data set. Therefore, records will be retained for up to five years for follow-on studies, provided each site agrees to this plan.

#### 8.3 Informed Consent/Assent and HIPAA Authorization

Waiver of informed consent has been granted for this retrospective chart review study as it meets the following criteria pursuant to 45 CRF 46.116(d):

- The research involves no more than minimal risk to the subjects.
- The waiver or alteration will not adversely affect the rights and welfare of the subjects.
- The research could not practicably be carried out without the waiver or alteration.

Waiver of HIPAA authorization has been granted as it meets the following criteria pursuant to 45 CFR 164.512(i)(1)(i)

- The use or disclosure of protected health information involves no more than a minimal risk to the privacy of individuals, based on, at least, the presence of the following elements:
  - o an adequate plan to protect the identifiers from improper use and disclosure;
  - o an adequate plan to destroy the identifiers at the earliest opportunity consistent with conduct of the research, unless there is a health or research justification for retaining the identifiers or such retention is otherwise required by law; and
  - adequate written assurances that the protected health information will not be reused or disclosed to any other person or entity, except as required by law, for authorized oversight of the research project, or for other research for which the use or disclosure of protected health information would be permitted by this subpart;
- The research could not practicably be conducted without the waiver or alteration; and
- The research could not practicably be conducted without access to and use of the protected health information.

# 9 APPENDIX: DATA TO BE OBTAINED FROM MASSACHUSETTS CARDIAC SURGICAL PROGRAMS

| Line | | | | STS 2.81<br>variable | STS 2.73<br>variable | STS 2.61<br>variable | STS 2.52<br>variable |
|---|---|---|---|---|---|---|---|
| number | Section | Variable text | STS variable names | numbers | numbers | numbers | numbers |
| 1 | | STS database version | | | | | |
| 2 | B. Demog | graphics | | | | | |
| 3 | | Patient Last Name | PatLName | 50 | 90 | 100 | 100 |
| 4 | | Patient First Name | PatFName | 55 | 100 | 110 | 110 |
| 5 | | Zip Code | PatZip | 105 | 210 | 180 | 180 |
| 6 | | Medical Record Number | MedRecN | 85 | 170 | 170 | 170 |
| 7 | | Date of Birth | DOB | 65 | 130 | 130 | 130 |
| 8 | | Gender | Gender | 75 | 150 | 150 | 150 |
| 9 | | Race | Race | - | - | 190 | 190 |
| 10 | | Race | RaceDocumented | 150 | - | - | - |
| 11 | | RaceCaucasian | RaceCaucasian | 155 | 290 | 191 | - |
| 12 | | RaceBlack | RaceBlack | 160 | 300 | 192 | - |
| 13 | | RaceAsian | RaceAsian | 165 | 310 | 193 | - |
| 14 | | RaceNativeAm | RaceNativeAm | 170 | 320 | 194 | - |
| 15 | | RacNativePacific | RacNativePacific | 175 | 330 | 195 | - |
| 16 | | RaceOther | RaceOther | 180 | 340 | 196 | - |
| 17 | | Ethnicity | Ethnicity | 185 | 350 | 199 | - |
| 18 | C. Hospi | talization | | | | | |
| 19 | | Hospital Name | HospName | 205 | 380 | 220 | 220 |
| 20 | | Date of Surgery | SurgDt | 310 | 610 | 260 | 260 |
| 21 | | Date of Discharge | DischDt | 315 | 620 | 270 | 270 |
| 22 | | Payor | PayorGov | 225 | 420 | 247 | - |
| 23 | | Payor | PayorComm | 275 | 510 | 254 | - |
| 24 | | Payor | PayorHMO | 280 | 520 | 255 | - |
| 25 | D. Risk Fa | actors | | | | | |
| 26 | | Height | HeightCm | 330 | 640 | 360 | 360 |
| 27 | | Weight | WeightKg | 335 | 630 | 350 | 350 |
| 28 | | Diabetes | Diabetes | 360 | 780 | 400 | 400 |

| 29 | Diabetes - control | DiabCtrl | 365 | 790 | 410 | 410 |
|---|---|---|---|---|---|---|
| 30 | Dyslipidemia | Dyslip | 370 | 800 | 420 | 420 |
| 31 | Dialysis | Dialysis | 375 | 810 | 450 | 450 |
| 32 | Hypertension | Hypertn | 380 | 820 | 460 | 460 |
| 33 | Smoker | TobaccoUse | 400 | - | - | - |
| 34 | Smoker | CigSmoker | - | 650 | 370 | 370 |
| 35 | Smoker | SmokCurr | - | 660 | - | - |
| 36 | Chronic Lung Disease | ChrLungD | 405 | 860 | 510 | 510 |
| 37 | Sleep Apnea | SlpApn | 460 | 950 | - | - |
| 38 | Alcohol Use | Alcohol | 480 | 1131 | - | - |
| | Peripheral Artery | | | | | |
| 39 | Disease | PVD | 505 | 980 | 530 | 530 |
| 40 | Cerebrovascular disease | CVD | 525 | 1010 | 540 | 540 |
| 41 | Prior CVA | CVA | 530 | 1020 | 470 | 470 |
| 42 | Prior CVA-When | CVAWhen | 535 | 1030 | 480 | 480 |
| 43 | CVD TIA | CVDTIA | 540 | 1050 | 540 | 540 |
| 44 | CVD Carotid stenosis | CVDCarSten | 545 | 1070 | 550 | 550 |
| 45 | Right carotid disease | CVDStenRt | 550 | 1071 | - | - |
| 46 | Left carotid disease | CVDStenLft | 555 | 1072 | - | - |
| 47 | Priot carotid surgery | CVDPCarSurg | 560 | 1080 | - | - |
| 48 | WBC Count | WBC | 565 | 690 | - | - |
| 49 | Last Creatinine | CreatLst | 585 | 750 | 430 | 430 |
| 50 | Infectious endocarditis | InfEndo | 385 | 830 | 490 | 490 |
| 51 | E. Previous Cardiac Interventions | | | | | |
| | Previous Cardiac | | | | | |
| 52 | Interventions | PrCVInt | 665 | 1200 | 570 | 570 |
| 53 | Previous CABG | PrCAB | 670 | 1215 | 600 | 600 |
| 54 | Previous Valve | PrValve | 675 | 1216 | 610 | 610 |
| | Previous valve surgery | | | | | |
| 55 | type 1 | PrValveProc1 | 695 | - | - | - |
| | Previous valve surgery | | | | | |
| 56 | type 2 | PrValveProc2 | 700 | - | - | - |
| | Other Previous Cardiac | | | | | |
| 57 | Interventions | POC | 805 | - | 620 | 620 |

| | Other previous cardiac | | | | | |
|----|--------------------------|--------------------|-----|------|-----|-----|
| 58 | intervention 1 | POCInt1 | 810 | - | - | - |
| | Other previous cardiac | | | | | |
| 59 | intervention 2 | POCInt2 | 815 | - | - | - |
| | Other previous cardiac | | | | | |
| 60 | intervention 3 | POCInt3 | 820 | - | - | - |
| | Previous carotid artery | | | | | |
| 61 | surgery | CVDPCarSurg (1080) | - | 1080 | 557 | 557 |
| 62 | Previous ICD | Procaicd | - | 1460 | 630 | 630 |
| 63 | Previous Pacemaker | PrOCPace | - | 1470 | 640 | 640 |
| | Previous arrhythmia | | | | | |
| 64 | surgery | POArr | - | 1445 | - | - |
| 65 | Previous other cardiac | PrOthCar | - | 1440 | - | - |
| 66 | Previous congenital | PrOthCongen | - | 1450 | 621 | - |
| | Previous Aortic Valve | | | | | |
| 67 | Replacement - Surgical | PrevProcAVReplace | - | 1220 | - | - |
| | Previous Aortic Valve | | | | | |
| 68 | Repair - Surgical | PrevProcAVRepair | - | 1230 | - | - |
| | Previous Mitral Valve | | | | | |
| 69 | Replacement - Surgical | PrevProcMVReplace | - | 1240 | - | - |
| | Previous Mitral Valve | | | | | |
| 70 | Repair - Surgical | PrevProcMVRepair | - | 1250 | - | - |
| | Previous Tricuspid Valve | | | | | |
| 71 | Replacement - Surgical | PrevProcTVReplace | - | 1260 | - | - |
| | Previous Tricuspid Valve | | | | | |
| 72 | Repair - Surgical | PrevProcTVRepair | - | 1270 | - | - |
| | Previous Pulmonic Valve | | | | | |
| | Repair / Replacement - | | | | | |
| 73 | Surgical | PrevProcPV | - | 1280 | - | - |
| | Previous Aortic Valve | | | | | |
| 74 | Balloon Valvuloplasty | PrevProcAVBall | - | 1285 | - | - |
| | Previous Mitral Valve | | | | | |
| 75 | Balloon Valvuloplasty | PrevProcMVBall | - | 1290 | - | - |
| 76 | Previous Transcatheter | PrevProcTCVRep | - | 1300 | - | - |

| | Valve Replacement | | | | | |
|---|---|---|---|---|---|---|
| | Previous Percutaneous | PrevProcPercVRepai | | | | |
| 77 | Valve Repair | r | - | 1310 | - | - |
| 78 | F. Preoperative Cardiac Status | | | | | |
| 79 | Previous MI | PrevMI | 885 | 1540 | 750 | 750 |
| 80 | Previous MI - when | MIWhen | 890 | 1550 | 760 | 760 |
| 81 | Prior Heart Failure | PriorHF | 920 | 1590 | 770 | 770 |
| 82 | History of Arrhythmia | Arrhythmia | 945 | - | 840 | 840 |
| 83 | History of Arrhythmia | ArrhythWhen | - | 1650 | - | - |
| 84 | VT/VF | ArrhyVtach | - | 1660 | 851 | - |
| | | ArrhyVtachSicSinSyn | | | | |
| 85 | Sick sinus syndrome | ; | - | 1680 | - | - |
| 86 | Third degree heart block | ArrhyTHB | - | 1690 | 852 | - |
| | Second degree heart | | | | | |
| 87 | block | ArrhyVtachHrtBlk | - | 1670 | - | - |
| 88 | VT/VF | ArrhythVV | 950 | - | - | - |
| 89 | Sick sinus syndrome | ArrhythSSS | 955 | - | - | - |
| 90 | Atrial Flutter | ArrhythAFlutter | 960 | - | - | - |
| | Second degree heart | | | | | |
| 91 | block | ArrhythSecond | 965 | - | - | - |
| 92 | Third degree heart block | ArrhythThird | 970 | - | - | - |
| 93 | Paced rhythm | ArrhythPPaced | 975 | - | - | - |
| 94 | Afib/Aflutter | ArrhythAFib | 980 | 1700 | 853 | - |
| 95 | Type of Atrial Fibrillation | ArrhyTyp | - | - | 850 | 850 |
| | Duration of Atrial | | | | | |
| 96 | Fibrillation | ArrythAFibDur | 985 | - | - | - |
| 97 | Type of Atrial Fibrillation | ArrythAFibTy | - | 1701 | - | - |
| 98 | G. Preoperative Medications | | | | | |
| 99 | ACE inhibitor Use | MedACEI48 | 1020 | 1730 | 900 | 900 |
| 100 | Anticoagulant Use | MedACoag | 1040 | 1750 | 940 | 940 |
| 101 | Amiodarone Use | MedAmiodarone | 1035 | - | - | - |
| 102 | Aspirin Use | MedASA | 1055 | 1820 | 990 | 990 |
| 103 | B-blockers <24 hours | MedBeta | 1060 | 1710 | 890 | 890 |
| 104 | B-blockers >2 weeks | MedBetaTher | 1065 | - | - | - |

| | | Calcium Channel | | | | | |
|---|---|---|---|---|---|---|---|
| 105 | | Blocker | MedCChanTher | 1070 | - | - | - |
| | | Preoperative | | | | | |
| 106 | | Antiarrhythmics | MedAArrhy | - | 1770 | - | - |
| 107 | | Coumadin | MedCoum | 1075 | 1780 | 950 | 950 |
| 108 | H. Hemo | odynamics Cath | | | | | |
| | | Number of Diseased | | | | | |
| 109 | | Vessels | NumDisV | 1170 | 1930 | 1050 | 1050 |
| 110 | | LV ejection fraction | HDEF | 1545 | 1960 | 1080 | 1080 |
| 111 | | Aortic Insufficiency | VDInsufA | 1590 | 2155 | 1170 | 1170 |
| 112 | | Aortic Stenosis | VDStenA | 1600 | 2152 | 1120 | 1120 |
| 113 | | Aortic Valve Area | VDAoVA | 1610 | 2153 | - | - |
| | | Aortic Valve Mean | | | | | |
| 114 | | Gradient | VDGradA | 1615 | 2154 | 1130 | 1130 |
| 115 | | Mitral Insufficiency | VDInsufM | 1680 | 2270 | 1180 | 1180 |
| 116 | | Mitral Stenosis | VDStenM | 1690 | 2240 | 1140 | 1140 |
| | | Mitral Valve Mean | | | | | |
| 117 | | Gradient | VDGradM | 1705 | 2260 | 1180 | 1180 |
| 118 | | Tricuspid Insufficiency | VDInsufT | 1775 | 2320 | 1190 | 1190 |
| 119 | | Tricuspid Stenosis | VDStenT | 1785 | 2300 | 1150 | 1150 |
| 120 | | Pulmonary Insufficiency | VDInsufP | 1820 | 2340 | 1200 | 1200 |
| 121 | | Pulmonary Stenosis | VDStenP | 1840 | 2330 | 1160 | 1160 |
| 122 | I. Opera | tive (with sections J, K, L and | d M) | | | | |
| 123 | | AF procedure | AFibProc | 2145 | - | 2470 | 2470 |
| 124 | | Afib epicardial lesions | OCarAFibEpLes | 4070 | - | - | - |
| 125 | | Afib intracardiac lesions | OCarAFibIntraLes | 4105 | - | - | - |
| 126 | | Aortic Arch | AortProcTotArch | 4355 | - | - | - |
| 127 | | Aortic Arch | ONCArch | - | - | 2530 | 2530 |
| 128 | | Aortic Arch | ONCArch | - | 5480 | - | - |
| 129 | | Aortic Hemi-arch | AortProcHemi | 4350 | - | - | - |
| 130 | | Aortic Procedure | AortProc | 2150 | - | - | - |
| 131 | | Aortic Procedure | OpAortic | - | - | 1630 | 1630 |
| 132 | | Aortic Procedure Type | OCAoProcType | - | 5471 | - | - |
| 133 | | Aortic Root | AortProcRoot | 4340 | - | - | - |

| 134 | Aortic Root | ONCAoRt | - | 5473 | - | - |
|---|---|---|---|---|---|---|
| 135 | Aortic Valve Procedure | VSAVPr | - | 4280 | - | - |
| 136 | Aortic Valve Surgery | VSAV | 3390 | 4270 | - | - |
| | Arrhythmia Correction | | | | | |
| 137 | Surgery | OCarACD | - | 5400 | - | - |
| | Arrhythmia Correction | | | | | |
| 138 | Surgery Lead Extraction | OCarACDLI | - | 5410 | - | - |
| 139 | Arrythmia device | OCarACD | 4085 | 5400 | 2450 | 2450 |
| 140 | Ascending Aorta | AortProcAsc | 4345 | - | - | - |
| 141 | Ascending Aorta | ONCAsc | - | - | 2520 | 2520 |
| 142 | Ascending Aorta | ONCAsc | - | 5474 | - | - |
| 143 | ASD-PFO repair | OCarASD | | 5240 | - | - |
| 144 | ASD-PFO repair | OCarASDPFO | 4075 | - | - | - |
| | Atrial Appendage | | | | | |
| 145 | Procedure | OCarAAProc | 4080 | - | 2480 | 2480 |
| | Atrial Fibrillation | | | | | |
| 146 | Ablation Procedure | OCarAFibAProc | - | 5465 | - | - |
| | Atrial Fibrillation Surgical | | | | | |
| 147 | Procedure | OCarAFibSur | - | 5450 | - | - |
| 148 | CABG performed | ОрСАВ | 2120 | 2437 | 1280 | 1280 |
| 149 | Cardiac trauma | OCarTrma | 4153 | 5380 | 2430 | 2430 |
| 150 | Cardiac Tumor | OCTumor | 4150 | 5530 | - | - |
| 151 | Congenital heart surgery | OCarCong | 4162 | 5300 | 2410 | 2410 |
| 152 | Congenital procedure 1 | OCarCongProc1 | 4515 | 5340 | - | - |
| 153 | Congenital procedure 2 | OCarCongProc2 | 4520 | 5350 | - | - |
| 154 | Congenital procedure 3 | OCarCongProc3 | 4525 | 5360 | - | - |
| 155 | CPB time | PerfusTm | 2400 | 2770 | 1380 | 1380 |
| 156 | CPB utilization | CPBCmb | - | 2470 | 1360 | 1360 |
| 157 | CPB utilization | CPBUtil | 2325 | 2740 | 1350 | 1350 |
| 158 | Emergency Operation | Status | 1975 | 2390 | 1240 | 1240 |
| 159 | Heart transplant | OCarCrTx | 4152 | 5390 | 2440 | 2440 |
| 160 | Lead extraction | OCarACDLE | 4120 | - | - | - |
| 161 | Lead Insertion | OCarLeadInsert | 4090 | - | - | - |
| 162 | Left Atrial Appendage | OCarAFibSurLAA | - | 5452 | - | - |

| | Obliterated | | | | | |
|-----|-------------------------|-----------------|------|------|------|------|
| 163 | LV aneurysm repair | OCarLVA | 4125 | 5220 | 2360 | 2360 |
| 164 | Mitral Procedure | OpMitral | - | - | 1640 | 1640 |
| 165 | Mitral Valve Procedure | VSMVPr | - | 4352 | - | - |
| 166 | Mitral Valve Surgery | VSMV | 3495 | 4351 | - | - |
| | Number of anastomoses | | | | | |
| 167 | with arterial conduits | DistArt | 2625 | 3190 | 1520 | 1520 |
| | Number of anastomoses | | | | | |
| 168 | with venous conduits | DistVein | 2630 | 3220 | 1530 | 1530 |
| | Other Cardiac | | | | | |
| 169 | Procedure | OpOCard | 2140 | 2490 | 1310 | 1310 |
| 170 | Previous VAD | PrevVAD | 3790 | 4760 | 1920 | 1920 |
| | Pulmonary | | | | | |
| | thromboendarterectom | | | | | |
| 171 | у | OCPulThromDis | 4130 | 5540 | - | - |
| | Pulmonic Valve | | | | | |
| 172 | Procedure | OpPulm | - | 4560 | - | - |
| 173 | Pulmonic Valve Surgery | VSPV | 3685 | - | 1660 | 1660 |
| 174 | Reop surgery | Incidenc | 1970 | 2380 | 560 | 560 |
| | Subaortic stenosis | | | | | |
| 175 | reseaction | OCarSubaStenRes | 4135 | - | - | - |
| | Subaortic stenosis | | | | | |
| 176 | reseaction | ResectSubA | - | 4311 | - | - |
| | Surgical Procedure | | | | | |
| 177 | Location | OCarAFibSurLoc | - | 5451 | - | - |
| | Surgical ventricular | | | | | |
| 178 | restoration | OCarSVR | 4145 | 5290 | 2400 | 2400 |
| 179 | TMR | OCarLasr | 4100 | 5370 | 2420 | 2420 |
| | Tricuspid Valve | | | | | |
| 180 | Procedure | OpTricus | - | 4500 | - | - |
| 181 | Tricuspid Valve Surgery | VSTV | 3640 | - | 1650 | 1650 |
| 182 | VAD implant type | VImpTy | - | 4850 | - | - |
| 183 | VAD implanted | VADImp | 3840 | - | 2030 | 2030 |
| 184 | VAD Implanted or | VADProc | 2130 | 2480 | - | - |

| | | Removed | | | | | |
|---|---|---|---|---|---|---|---|
| 185 | | Valve Surgery | OpValve | 2125 | 2440 | 1290 | 1290 |
| 186 | | VSD repair | OCarVSD | 4155 | 5230 | 2370 | 2370 |
| 187 | N. Other | Non-Cardiac Procedures | | | | | |
| 188 | | Carotid endarterectomy | ONCCarEn | 4530 | 5560 | 2570 | 2570 |
| 189 | P. Posto | perative Events | | | | | |
| 190 | | Postop stroke | CNStrokP | 4810 | 6030 | 2630 | 2630 |
| 191 | | Postop TIA | CNStrokTTIA | 4815 | 6040 | 2840 | 2840 |
| 192 | | Atrial Fibrillation | COAtFib | 4930 | 6330 | 2990 | 2990 |
| 193 | | Reop for bleeding | COpReBld | 4755 | 5760 | 2720 | 2720 |
| | | Postop pacemaker | | | | | |
| 194 | | insertion | CRhythmDis | 4900 | 6270 | - | - |
| 195 | Q. Morta | ality | | | | | |
| 196 | | Mortality | Mortality | 5005 | 6360 | 3020 | 3020 |
| 197 | | Date of Death | MtDate | 5030 | 6400 | 3060 | 3060 |
| 198 | | Primary cause of death | MtCause | 5040 | 6420 | 3080 | 3080 |
| 199 | R. Discha | arge (with Section S) | | | | | |
| 200 | | Aspirin | DCASA | 5060 | 6460 | 3120 | 3120 |
| 201 | | Warfarin | DCCoum | 5085 | 6510 | 3180 | 3180 |
| 202 | | Antiarrythmic | DCAArhy | - | 6440 | 3100 | 3100 |
| 203 | | Antiarrythmic name | DCAArMN | - | - | 3110 | 3110 |
| 204 | | Readmission | Readm30 | - | 6550 | 3220 | 3220 |
| | | Primary readmission | | | | | |
| 205 | | reason | ReadmRsn | - | 6560 | 3230 | 3230 |
| 206 | | Amiodarone | DCAmiodarone | 5110 | - | - | - |
| 207 | | Beta-blocker | DCBeta | 5105 | 6480 | 3140 | 3140 |
| 208 | | Discharge location | DisLoctn | 5045 | 6520 | 3190 | 3190 |

#### 10 APPENDIX: CHIA-SOURCED VARIABLE DEFINITIONS AND ABSTRACTION

We will create a subset of cardiac surgery patients using all three CHIA databases to maximize the chance of finding a matching cardiac surgery record in RPDR. UHINs for the cardiac surgery cases are identified in the inpatient database where at least one of 15 procedure codes or principal procedure contains an ICD9-CM code for cardiac surgery (3610-3619). The following lists the minimum set of fields needed to complete the merge.

- a. MDPHHospNum: MDPH hospital number determined from all hospital IDs in the case mix data
- b. AdmitDt: Admission date to hospital
- c. ProcDates: Possible dates for cardiac surgical procedure (15 in inpatient, 3 in OOR data)
- d. ProcedureCodes: ICD-9-CM and CPT (OOR only) codes for cardiac surgery records (only 3 ICD-9-CM in OOR data)
- e. PrincipalProcDate: Date for principal procedure (OOR only)
- f. PrincipalProcedure: ICD9-CM code for PCI and CABG records
- g. Diagnosis Codes: Diagnosis and DRG codes for conditions
- h. DischDate: Discharge date from hospital
- RecordType20ID: CHIA Record Id Control Number
- j. UHIN Unique patient identifier from CHIA
- k. DOB: Patient date of birth submitted by hospital
- I. MedicalRecordNum: Hospital patient medical record number
- m. Gender: Patient gender

# 11 APPENDIX: PROPOSED TIMELINE

| Activity | Jan-Feb<br>2018 | Feb-Mar<br>2018 | Apr-May<br>2018 | May-Jul<br>2018 | Jul-Sep<br>2018 | Sep-Oct<br>2018 | Oct-Nov<br>2018 |
|---|---|---|---|---|---|---|---|
| Study design | | | | | | | |
| IRB and DUA approval | | | | | | | |
| Data submission and | | | | | | | |
| merging at CHIA | | | | | | | |
| Data cleaning and | | | | | | | |
| analysis | | | | | | | |
| Analysis write-up and | | | | | | | |
| first circulation | | | | | | | |
| Paper preparation and | | | | | | | |
| second circulation | | | | | | | |
| Paper submission | | | | | | | |

#### 12 APPENDIX: SHELL TABLES AND FIGURES

#### 12.1 Tables

- Table 1: Characteristics of the study participants.
- Table 2: Comparison of characteristics of patients with post-discharge atrial fibrillation and those patients who did not have post-discharge atrial fibrillation
- Table 3: Time-adjusted risk of post-discharge atrial fibrillation
- Table 4: Time-adjusted risk of post-discharge stroke
- Table 5: Time-adjusted risk of post-discharge mortality

#### 12.2 Figures

- Figure 1: CONSORT diagram
- Figure 2: Time course of the occurrence of post-discharge AF
- Figure 3: Time course of the occurrence of post-discharge stroke stratified by occurrence of post-discharge AF
- Figure 4: Time course of the occurrence of post-discharge mortality stratified by occurrence of post-discharge AF

**Table 1:** Characteristics of the study participants. Data are reported as number and percentage, or median and 10-90% quantiles, as appropriate

CSP = Cardiac surgical program

CHIA = Center for Health Information and Analysis

| | Patient characteristic | Data source | Source variable |
|---|---|---|---|
| 0 | Demographics | | |
| 1 | Age at surgery (years; N/%) | CSP | Calculated |
| 2 | <50 | | SurgDt - DOB |
| 3 | 50-59 | | |
| 4 | 60-69 | | |
| 5 | 70-79 | | |
| 6 | ≥80 | | |
| 7 | Gender (Male; N/%) | CSP | Gender |
| 8 | Race (Caucasian; N/%) | CSP | RaceCaucasian |
| 9 | Ethnicity | CSP | Ethnicity |
| 10 | Height (cm; mean/SD) | CSP | HeightCm |
| 11 | Weight (kg; mean/SD) | CSP | WeightKg |
| 12 | BMI (kg/m2; N/%) | CSP | Calculated |
| 13 | <20 | | |
| 14 | 20-24.9 | | |
| 15 | 25-29.9 | | |
| 16 | 30-34.9 | | |
| 17 | ≥35 | | |
| 18 | Payor | | |
| 19 | Government | CSP | PayorGov |
| 20 | Commercial | CSP | PayorComm |
| 21 | НМО | CSP | PayorHMO |
| 22 | Prior Medical History | | ArrhythAFib, ArrythAFibDur, ArrythAFibTy |
| 23 | Atrial fibrillation | CSP and CHIA | ArrhythAFlutter |
| 24 | Atrial flutter | CSP and CHIA | Armythariated |
| 25 | History of arrhythmia | CSP and CHIA | |
| 26 | Heart block or sick sinus syndrome | CSP and CHIA | ArrhyVtachSicSinSyn, ArrhyTHB, ArrhyVtachHrtBlk, |
| | | | ArrhythSSS |

| 27 | VT/VF | CSP and CHIA | ArrhyVtach, ArrhythVV |
|---|---|---|---|
| 28 | Smoker past or current | CSP | TobaccoUse, CigSmoker, SmokCurr |
| 29 | COPD | CSP | ChrLungD |
| 30 | Diabetes | CSP | Diabetes, DiabCtrl |
| 31 | NIDDM | | |
| 32 | IDDM | | |
| 33 | Dyslipidemia | CSP | Dyslip |
| 35 | Dialysis | CSP | Dialysis |
| 36 | Hypertension | CSP | Hypertn |
| 37 | Peripheral vascular disease | CSP | PVD |
| 38 | Sleep apnea | CSP | SlpApn |
| 39 | Alcohol use | CSP | Alcohol |
| 40 | Cerebrovascular disease | CSP | CVD |
| 41 | Prior CVA | CSP | CVA, CVAWhen |
| 42 | TIA | CSP | CVDTIA |
| 43 | Carotid Stenosis | CSP | CVDCarSten |
| 44 | Prior carotid surgery | CSP | CVDPCarSurg |
| 45 | | | |
| 46 | Medications | | |
| 47 | ACEI/ARB | CSP | MedACEI48 |
| 48 | Anticoagulant or anti-platelet drug | CSP | MedACoag |
| 49 | Amiodarone | CSP | MedAmiodarone |
| 50 | Aspirin | CSP | MEDASA |
| 51 | Beta blocker | CSP | MedBeta |
| 52 | Calcium channel blocker | CSP | MedCChanTher |
| 53 | Antiarrythmic | CSP | MedAArry |
| 54 | Coumadin | CSP | MedCoum |
| 55 | | | |
| 56 | Prior Cardiac Status | | |
| 57 | Heart failure | | PriorHF |
| 58 | Prior MI | | PrevMI, MIWhen |
| 59 | Past | | |
| 60 | Recent | | |
| 61 | Prior CABG surgery | CSP | PrCAB |

| 62 | Prior mitral valve surgery | CSP | PrValveProc1, PrValveProc2, PrevProcMVReplace, |
|---|---|---|---|
| | <b>0</b> , | | PreProcMVRepair |
| 63 | Prior other valve surgery | CSP | PrValveProc1, PrValveProc2, PrevProcAVReplace, |
| | 3 , | | PrevProcAVRepair , PrevProcTVReplace , |
| | | | PrevProcTVRepair , PrevProcPV , PrevProcAVBall , |
| | | | PrevProcMVBall , PrevProcTCVRep , |
| | | | PrevProcPercVRepair |
| 64 | Other cardiac surgery | CSP | PrOthCar, PrOthCongen, POC, POCInt1, POCInt2, |
| 01 | | | POCInt3 |
| 65 | Prior ICD placement | CSP | Procaicd |
| 66 | Prior pacemaker placement | CSP | PrOCPace |
| 67 | Prior arrhythmia surgery | CSP | POArr |
| 69 | The anniquence of geny | | 1.67.11 |
| 70 | Preoperative laboratory testing | | |
| 77 | White cell count (10 <sup>6</sup> /dL) | CSP | WBC |
| 78 | Creatinine (mg/dL) | CSP | CreatLst |
| 79 | | | 5.53.25 |
| 80 | Preoperative Cardiac Imaging | | |
| 81 | Number of diseased coronary | CSP | NumDisV |
| | vessels | | |
| 82 | 0 | | |
| 83 | 1 | | |
| 82 | 2 | | |
| 83 | >=3 | | |
| 84 | LV Ejection fraction | CSP | HDEF |
| 85 | <30% | | |
| 86 | 30-54% | | |
| 87 | >=55% | | |
| 88 | Aortic stenosis | CSP | VDStenA |
| 89 | Aortic insufficiency | CSP | VDInsufA |
| 90 | Mitral stenosis | CSP | VDStenM |
| 91 | Mitral insufficiency | CSP | VDinsufM |
| 92 | Tricuspid valve disease | CSP | VDStenT, VDStenP |
| 93 | Pulmonary valve disease | CSP | VDStenP, VDinsufP |

| 94 | | | |
|---|---|---|---|
| 95 | Surgery | | |
| 96 | Year of operation | CSP | SurgDt |
| 97 | 2012 | | |
| 98 | 2013 | | |
| 99 | 2014 | | |
| 100 | 2015 | | |
| 101 | 2016 | | |
| 101 | CABG surgery | CSP | OpCAB |
| 102 | Number of conduits placed | CSP | DistArt + DistVein |
| 103 | 1 | | |
| 104 | 2 | | |
| 105 | >=3 | | |
| 106 | AVR surgery | CSP | VSAVPr, VSAV |
| 107 | MVR surgery | CSP | OpMitral, VSMVPr, VSMV |
| 108 | Other valve surgery | CSP | OpPulm, VSPV, OpTricus, VSTV |
| 109 | Ascending aortic surgery | CSP | A ort Proc Tot Arch, ON CArch, A ort Proc Hemi, A ort Proc , |
| | | | OpAortic, OCAoProcType, AortProcRoot, ONCAoRt, |
| | | | AortProcAsc, ONCAsc, ONCAsc |
| 110 | Other non-CABG, non valvular | CSP | OpOCard |
| | surgery | | |
| 111 | Atrial septal surgery | CSP | OCarASD, OCarASDPFO |
| 114 | Ventricular outflow tract surgery | CSP | OCarSubaStenRes , ResectSubA |
| 115 | Congenital heart surgery | | ${\sf OCarCong},{\sf OCarCongProc1},{\sf OCarCongProc2},$ |
| | | | OCarCongProc3 |
| 116 | Carotid endarterectomy | CSP | |
| 117 | Reoperation | CSP | Incidenc |
| 118 | Surgical urgency | CSP | Status |
| 119 | Elective | | |
| 120 | Urgent | | |
| 121 | Emergent | | |
| 122 | Postoperative duration (days) | CSP | DischDt - SurgDt |
| 123 | | | |
| 124 | Post-operative complications | | |

| 125 | Stroke | CSP and CHIA | CNStrokP |
|-----|------------------------------------|--------------|--------------|
| 126 | TIA | CSP and CHIA | CNStrokTTIA |
| 127 | Atrial fibrillation | CSP and CHIA | COAtFib |
| 128 | Reoperation for bleeding | CSP and CHIA | COpReBld |
| 129 | Pacemaker inserted | CSP and CHIA | CRythmDis |
| 130 | In-hospital atrial fibrillation | CSP | COAtFib |
| 131 | In-hospital atrial flutter | CSP | |
| 132 | | | |
| 133 | Discharge medications and devices | | |
| 134 | Aspirin | CSP and CHIA | DCASA |
| 135 | Warfarin | CSP and CHIA | DCCoum |
| 136 | Anti-platelet agent | CHIA | - |
| 137 | Beta blocker | CSP and CHIA | DCBeta |
| 138 | Amiodarone | CSP and CHIA | DCAmiodarone |
| 139 | | | |
| 140 | Post-discharge atrial fibrillation | | |
| 141 | Discharged in AF | CSP | |
| 142 | 1 - 30 days | CHIA | |
| 143 | 31 - 90 days | CHIA | |
| 144 | 91 - 182 days | CHIA | |
| 145 | 183 - 365 days | CHIA | |
| 146 | 1 - 2 years | CHIA | |
| 147 | 2 - 3 years | CHIA | |
| 148 | 3 – 4 years | CHIA | |
| 149 | 4 - 5 years | CHIA | |
| 150 | | | |
| 151 | Post-discharge stroke | CLUA | |
| 152 | 1 - 30 days | CHIA | |
| 154 | 31 - 90 days | CHIA | |
| 155 | 91 - 182 days | CHIA | |
| 156 | 183 - 365 days | CHIA | |
| 157 | 1 - 2 years | CHIA | |
| 158 | 2 - 3 years | CHIA | |
| 159 | 3 - 4 years | CHIA | |

| 160 | | 4 – 5 years | CHIA | |
|-----|------------------|-------------|------|-----------------------------|
| 161 | | | | |
| 162 | Mortality | | | |
| 163 | 30-day mortality | | CSP | Mortality and MortalityDate |
| 164 | 1-year mortality | | CSP | Mortality and MortalityDate |
| 165 | 5-year mortality | | CSP | Mortality and MortalityDate |

Table 2: Comparison of characteristics of patients with post-discharge atrial fibrillation and those patients who did not have post-discharge atrial fibrillation

Figure 1: CONSORT Diagram.

| Patients reported in local STS databases<br>Operations reported local STS databases |
|---|

Excluded after matching

- x,xxx patients
- x,xxx operations

#### Excluded after data review (N=x,xxx)

- Inclusion criterion not present
- Exclusion criterion present
- Covariate data not present
- Missing outcome

Eligible patients (N = xx,xxx)

CABG-only surgery (N = xx,xxx)

AVR +/- CABG surgery (N = xx,xxx)

MVR +/- AVR +/- CABG surgery (N = xx,xxx)

### 13 APPENDIX: STROBE CRITERIA

STROBE Statement—Checklist of items that should be included in reports of *cohort studies* 

| | Item<br>No | Recommendation |
|---|---|---|
| Title and abstract | 1 | (a) Indicate the study's design with a commonly used term in the title or the abstract |
| | | (b) Provide in the abstract an informative and balanced summary of what was done |
| | | and what was found |
| Introduction | | |
| Background/rationale | 2 | Explain the scientific background and rationale for the investigation being reported |
| Objectives | 3 | State specific objectives, including any prespecified hypotheses |
| Methods | | |
| Study design | 4 | Present key elements of study design early in the paper |
| Setting | 5 | Describe the setting, locations, and relevant dates, including periods of recruitment, |
| | | exposure, follow-up, and data collection |
| Participants | 6 | (a) Give the eligibility criteria, and the sources and methods of selection of |
| | | participants. Describe methods of follow-up |
| | | (b) For matched studies, give matching criteria and number of exposed and |
| | | unexposed |
| Variables | 7 | Clearly define all outcomes, exposures, predictors, potential confounders, and effect |
| | | modifiers. Give diagnostic criteria, if applicable |
| Data sources/ | 8* | For each variable of interest, give sources of data and details of methods of |
| measurement | | assessment (measurement). Describe comparability of assessment methods if there is |
| | | more than one group |
| Bias | 9 | Describe any efforts to address potential sources of bias |
| Study size | 10 | Explain how the study size was arrived at |
| Quantitative variables | 11 | Explain how quantitative variables were handled in the analyses. If applicable, |
| | | describe which groupings were chosen and why |
| Statistical methods | 12 | (a) Describe all statistical methods, including those used to control for confounding |
| | | (b) Describe any methods used to examine subgroups and interactions |
| | | (c) Explain how missing data were addressed |
| | | (d) If applicable, explain how loss to follow-up was addressed |
| | | (e) Describe any sensitivity analyses |
| Results | | |
| Participants | 13* | (a) Report numbers of individuals at each stage of study—eg numbers potentially |
| | | eligible, examined for eligibility, confirmed eligible, included in the study, |
| | | completing follow-up, and analysed |
| | | (b) Give reasons for non-participation at each stage |
| | | (c) Consider use of a flow diagram |
| Descriptive data | 14* | (a) Give characteristics of study participants (eg demographic, clinical, social) and |
| | | information on exposures and potential confounders |
| | | (b) Indicate number of participants with missing data for each variable of interest |
| | | (c) Summarise follow-up time (eg, average and total amount) |
| Outcome data | 15* | Report numbers of outcome events or summary measures over time |
| Main results | 16 | (a) Give unadjusted estimates and, if applicable, confounder-adjusted estimates and |
| | | their precision (eg, 95% confidence interval). Make clear which confounders were |
| | | adjusted for and why they were included |
| | | (b) Report category boundaries when continuous variables were categorized |
| | | (c) If relevant, consider translating estimates of relative risk into absolute risk for a |
| | | meaningful time period |

1

| Other analyses | 17 | Report other analyses done—eg analyses of subgroups and interactions, and sensitivity analyses |
|---|---|---|
| Discussion | | |
| Key results | 18 | Summarise key results with reference to study objectives |
| Limitations | 19 | Discuss limitations of the study, taking into account sources of potential bias or imprecision. Discuss both direction and magnitude of any potential bias |
| Interpretation | 20 | Give a cautious overall interpretation of results considering objectives, limitations, multiplicity of analyses, results from similar studies, and other relevant evidence |
| Generalisability | 21 | Discuss the generalisability (external validity) of the study results |
| Other information | | |
| Funding | 22 | Give the source of funding and the role of the funders for the present study and, if applicable, for the original study on which the present article is based |

<sup>\*</sup>Give information separately for exposed and unexposed groups.

Note: An Explanation and Elaboration article discusses each checklist item and gives methodological background and published examples of transparent reporting. The STROBE checklist is best used in conjunction with this article (freely available on the Web sites of PLoS Medicine at http://www.plosmedicine.org/, Annals of Internal Medicine at http://www.annals.org/, and Epidemiology at http://www.epidem.com/). Information on the STROBE Initiative is available at http://www.strobe-statement.org.

#### 14 APPENDIX: REFERENCES

- 1. Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the U.S. adult population. The American journal of cardiology 2013;112:1142-7.
- 2. Saxena A, Dinh DT, Reid CM, Smith JA, Shardey GC, Newcomb AE. Does preoperative atrial fibrillation portend a poorer prognosis in patients undergoing isolated aortic valve replacement? A multicentre Australian study. The Canadian journal of cardiology 2013;29:697-703.
- 3. Saxena A, Dinh D, Dimitriou J et al. Preoperative atrial fibrillation is an independent risk factor for mid-term mortality after concomitant aortic valve replacement and coronary artery bypass graft surgery. Interactive cardiovascular and thoracic surgery 2013;16:488-94.
- 4. Wang TK, Ramanathan T, Choi DH, Gamble G, Ruygrok P. Preoperative atrial fibrillation predicts mortality and morbidity after aortic valve replacement. Interactive cardiovascular and thoracic surgery 2014;19:218-22.
- 5. Kievisas M, Keturakis V, Vaitiekunas E, Dambrauskas L, Jankauskiene L, Kinduris S. Prognostic factors of atrial fibrillation following coronary artery bypass graft surgery. General thoracic and cardiovascular surgery 2017;65:566-574.
- 6. Fengsrud E, Englund A, Ahlsson A. Pre- and postoperative atrial fibrillation in CABG patients have similar prognostic impact. Scandinavian cardiovascular journal : SCJ 2017;51:21-27.
- 7. Levy F, Rusinaru D, Marechaux S, Charles V, Peltier M, Tribouilloy C. Determinants and prognosis of atrial fibrillation in patients with aortic stenosis. The American journal of cardiology 2015;116:1541-6.
- 8. Quader MA, McCarthy PM, Gillinov AM et al. Does preoperative atrial fibrillation reduce survival after coronary artery bypass grafting? The Annals of thoracic surgery 2004;77:1514-22; discussion 1522-4.
- 9. Attaran S, Saleh HZ, Shaw M, Ward A, Pullan M, Fabri BM. Does the outcome improve after radiofrequency ablation for atrial fibrillation in patients undergoing cardiac surgery? A propensity-matched comparison. European journal of cardio-thoracic surgery: official journal of the European Association for Cardio-thoracic Surgery 2012;41:806-10; discussion 810-1.
- 10. Ngaage DL, Schaff HV, Barnes SA et al. Prognostic implications of preoperative atrial fibrillation in patients undergoing aortic valve replacement: is there an argument for concomitant arrhythmia surgery? The Annals of thoracic surgery 2006;82:1392-9.
- 11. Saxena A, Virk SA, Bowman S, Bannon PG. Systematic review and meta-analysis on the impact of preoperative atrial fibrillation on short- and long-term outcomes after aortic valve replacement. The Journal of cardiovascular surgery 2017;58:943-950.
- 12. Ahlsson A, Fengsrud E, Bodin L, Englund A. Postoperative atrial fibrillation in patients undergoing aortocoronary bypass surgery carries an eightfold risk of future atrial fibrillation and a doubled cardiovascular mortality. European journal of cardio-thoracic surgery: official journal of the European Association for Cardio-thoracic Surgery 2010;37:1353-9.

- 13. Elahi M, Hadjinikolaou L, Galinanes M. Incidence and clinical consequences of atrial fibrillation within 1 year of first-time isolated coronary bypass surgery. Circulation 2003;108 Suppl 1:II207-12.
- 14. Pillarisetti J, Patel A, Bommana S et al. Atrial fibrillation following open heart surgery: long-term incidence and prognosis. Journal of interventional cardiac electrophysiology: an international journal of arrhythmias and pacing 2014;39:69-75.
- 15. El-Chami MF, Merchant FM, Smith P et al. Management of New-Onset Postoperative Atrial Fibrillation Utilizing Insertable Cardiac Monitor Technology to Observe Recurrence of AF (MONITOR-AF). Pacing and clinical electrophysiology: PACE 2016;39:1083-1089.
- 16. Lee R, McCarthy PM, Wang EC et al. Midterm survival in patients treated for atrial fibrillation: a propensity-matched comparison to patients without a history of atrial fibrillation. The Journal of thoracic and cardiovascular surgery 2012;143:1341-51; discussion 1350-1.
- 17. Lim E, Barlow CW, Hosseinpour AR et al. Influence of atrial fibrillation on outcome following mitral valve repair. Circulation 2001;104:159-63.
- 18. Magruder JT, Collica S, Belmustakov S et al. Predictors of Late-Onset Atrial Fibrillation Following Isolated Mitral Valve Repairs in Patients With Preserved Ejection Fraction. Journal of cardiac surgery 2016;31:486-92.
- 19. Mariscalco G, Klersy C, Zanobini M et al. Atrial fibrillation after isolated coronary surgery affects late survival. Circulation 2008;118:1612-8.
- 20. Horwich P, Buth KJ, Legare JF. New onset postoperative atrial fibrillation is associated with a long-term risk for stroke and death following cardiac surgery. Journal of cardiac surgery 2013;28:8-13.
- 21. Al-Atassi T, Kimmaliardjuk DM, Dagenais C, Bourke M, Lam BK, Rubens FD. Should We Ablate Atrial Fibrillation During Coronary Artery Bypass Grafting and Aortic Valve Replacement? The Annals of thoracic surgery 2017;104:515-522.
- 22. Elbadawi A, Ogunbayo GO, Elgendy IY et al. Impact of Left Atrial Appendage Exclusion on Cardiovascular Outcomes in Patients With Atrial Fibrillation Undergoing Coronary Artery Bypass Grafting (From the National Inpatient Sample Database). The American journal of cardiology 2017;120:953-958.
- 23. Endo D, Kato TS, Iwamura T et al. The impact of surgical left atrial appendage amputation/ligation on stroke prevention in patients undergoing off-pump coronary artery bypass grafting. Heart and vessels 2017;32:726-734.
- 24. Gillinov AM, Gelijns AC, Parides MK et al. Surgical ablation of atrial fibrillation during mitral-valve surgery. The New England journal of medicine 2015;372:1399-409.
- 25. Rankin JS, Lerner DJ, Braid-Forbes MJ, Ferguson MA, Badhwar V. One-year mortality and costs associated with surgical ablation for atrial fibrillation concomitant to coronary artery bypass grafting. European journal of cardio-thoracic surgery: official journal of the European Association for Cardio-thoracic Surgery 2017;52:471-477.
- 26. Abreu Filho CA, Lisboa LA, Dallan LA et al. Effectiveness of the maze procedure using cooled-tip radiofrequency ablation in patients with permanent atrial fibrillation and rheumatic mitral valve disease. Circulation 2005;112:120-5.
- 27. Blomstrom-Lundqvist C, Johansson B, Berglin E et al. A randomized double-blind study of epicardial left atrial cryoablation for permanent atrial fibrillation in patients undergoing mitral

- valve surgery: the SWEDish Multicentre Atrial Fibrillation study (SWEDMAF). European heart journal 2007;28:2902-8.
- 28. Chevalier P, Leizorovicz A, Maureira P et al. Left atrial radiofrequency ablation during mitral valve surgery: a prospective randomized multicentre study (SAFIR). Archives of cardiovascular diseases 2009;102:769-75.
- 29. Gillinov AM, Bhavani S, Blackstone EH et al. Surgery for permanent atrial fibrillation: impact of patient factors and lesion set. The Annals of thoracic surgery 2006;82:502-13; discussion 513-4.
- 30. Ad N, Holmes SD, Pritchard G, Shuman DJ. Association of operative risk with the outcome of concomitant Cox Maze procedure: a comparison of results across risk groups. The Journal of thoracic and cardiovascular surgery 2014;148:3027-33.
- 31. Damiano RJ, Jr., Lawrance CP, Saint LL et al. Detection of Atrial Fibrillation After Surgical Ablation: Conventional Versus Continuous Monitoring. The Annals of thoracic surgery 2016;101:42-7; discussion 47-8.
- 32. Melo J, Santiago T, Aguiar C et al. Surgery for atrial fibrillation in patients with mitral valve disease: results at five years from the International Registry of Atrial Fibrillation Surgery. The Journal of thoracic and cardiovascular surgery 2008;135:863-9.
- 33. Badhwar V, Rankin JS, Ad N et al. Surgical Ablation of Atrial Fibrillation in the United States: Trends and Propensity Matched Outcomes. The Annals of thoracic surgery 2017;104:493-500.
- 34. Ad N, Barnett S, Lefrak EA et al. Impact of follow-up on the success rate of the cryosurgical maze procedure in patients with rheumatic heart disease and enlarged atria. The Journal of thoracic and cardiovascular surgery 2006;131:1073-9.
- 35. Gammie JS, Haddad M, Milford-Beland S et al. Atrial fibrillation correction surgery: lessons from the Society of Thoracic Surgeons National Cardiac Database. The Annals of thoracic surgery 2008;85:909-14.
- 36. Calkins H, Kuck KH, Cappato R et al. 2012 HRS/EHRA/ECAS expert consensus statement on catheter and surgical ablation of atrial fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design: a report of the Heart Rhythm Society (HRS) Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. Developed in partnership with the European Heart Rhythm Association (EHRA), a registered branch of the European Society of Cardiology (ESC) and the European Cardiac Arrhythmia Society (ECAS); and in collaboration with the American College of Cardiology (ACC), American Heart Association (AHA), the Asia Pacific Heart Rhythm Society (APHRS), and the Society of Thoracic Surgeons (STS). Endorsed by the governing bodies of the American College of Cardiology Foundation, the American Heart Association, the European Cardiac Arrhythmia Society, the European Heart Rhythm Association, the Society of Thoracic Surgeons, the Asia Pacific Heart Rhythm Society, and the Heart Rhythm Society. Heart rhythm 2012;9:632-696 e21.
- 37. January CT, Wann LS, Alpert JS et al. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation 2014;130:2071-104.
- 38. Ad N, Cheng DC, Martin J et al. Surgical Ablation for Atrial Fibrillation in Cardiac Surgery: A Consensus Statement of the International Society of Minimally Invasive Cardiothoracic Surgery (ISMICS) 2009. Innovations (Philadelphia, Pa) 2010;5:74-83.

- 39. Badhwar V, Rankin JS, Damiano RJ, Jr. et al. The Society of Thoracic Surgeons 2017 Clinical Practice Guidelines for the Surgical Treatment of Atrial Fibrillation. The Annals of thoracic surgery 2017;103:329-341.
- 40. Ad N, Henry L, Hunt S, Holmes SD. Do we increase the operative risk by adding the Cox Maze III procedure to aortic valve replacement and coronary artery bypass surgery? The Journal of thoracic and cardiovascular surgery 2012;143:936-44.
- 41. Ad N, Cox JL. The Maze procedure for the treatment of atrial fibrillation: a minimally invasive approach. Journal of cardiac surgery 2004;19:196-200.
- 42. Worku B, Pak SW, Cheema F et al. Incidence and predictors of pacemaker placement after surgical ablation for atrial fibrillation. The Annals of thoracic surgery 2011;92:2085-9.
- 43. Shih T, Paone G, Theurer PF, McDonald D, Shahian DM, Prager RL. The Society of Thoracic Surgeons Adult Cardiac Surgery Database Version 2.73: More Is Better. The Annals of thoracic surgery 2015;100:516-21.
- 44. Jacobs JP, Shahian DM, He X et al. Penetration, Completeness, and Representativeness of The Society of Thoracic Surgeons Adult Cardiac Surgery Database. The Annals of thoracic surgery 2016;101:33-41; discussion 41.
- 45. Richardson DB, Laurier D, Schubauer-Berigan MK, Tchetgen Tchetgen E, Cole SR. Assessment and indirect adjustment for confounding by smoking in cohort studies using relative hazards models. Am J Epidemiol 2014;180:933-40.
- 46. VanderWeele TJ, Ding P. Sensitivity Analysis in Observational Research: Introducing the E-Value. Ann Intern Med 2017;167:268-274.
- 47. Amorim LD, Cai J. Modelling recurrent events: a tutorial for analysis in epidemiology. Int J Epidemiol 2015;44:324-33.
- 48. Schafer JL. Multiple imputation: a primer. Statistical methods in medical research 1999;8:3-15.
- 49. Schafer JL, Graham JW. Missing data: our view of the state of the art. Psychological methods 2002;7:147-77.
- 50. Vesin A, Azoulay E, Ruckly S et al. Reporting and handling missing values in clinical studies in intensive care units. Intensive care medicine 2013;39:1396-404.
- 51. Vickers AJ, Altman DG. Statistics notes: missing outcomes in randomised trials. BMJ (Clinical research ed) 2013;346:f3438.